CLINICAL TRIAL: NCT04343534
Title: Online Trial Examining Validity and Reliability of the Shared Decision Making Process Survey in Adults With Depression
Brief Title: Examining Validity and Reliability of the Shared Decision Making Process Survey in Adults With Depression
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Karen Sepucha, Director of the Health Decision Sciences Center, Massachusetts General Hospital
Other Study IDs: 2019P001434-2
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: Depression
Keywords: shared decision making
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Original Shared Decision Making Process scale: Patients receive the original version of the Shared Decision Making Process scale.
- Revised Shared Decision Making Process scale: This group completes a new version of the scale with different wording for several items.

SUMMARY:
The purpose of this study is to test two differently worded versions of the Shared Decision Making Process scale in a sample of adults who have recently made a decision about treatment of depression. The main goals are to gather evidence of reliability, to test whether the generic version has similar psychometric performance to the original, and to extend generalizability of the findings to younger adults.

DETAILED DESCRIPTION:
The purpose of this study is to test two differently worded versions of the Shared Decision Making Process scale in a sample of adults who have recently made a decision about treatment of depression. The main goals are to gather evidence of psychometric performance of the scale, compare performance of different wording for items, and to extend generalizability of the findings to younger adults.

Subjects are randomly assigned to one of the two versions of the Shared Decision Making Process scale and complete a set of measures regarding their experiences with decision making for depression, demographics, and health status. A subset of respondents will complete the Shared Decision Making Process scale and selected other items again 1 week later to examine short term test-retest reliability.

Staff will work with a national sampling firm to recruit subjects and obtain 500 responses to the baseline survey (n=250 for each version) and a subset will complete a retest survey (n=200; 50 from each age and survey type group). Eligible subjects are adults aged 18-75 who talked with a health care provider about treatment for depression in the preceding 12 months. The sample is not a national probability sample; however, the recruitment efforts will ensure about 50% of respondents aged 18-39 and 50% aged 40-75, and to ensure at least 25% of the sample is racial/ethnic minorities (Black or African American, Asian, Hispanic or Latino).

The investigators will examine validity and reliability of the different versions. The sample size was determined to ensure sufficient power to detect differences in key subgroups, including age (younger adults vs. older adults) and version (A vs. B). To detect a difference of about 0.33 standard deviations at 0.05 significance with 80% power would require 125 per group.

ELIGIBILITY:
Inclusion Criteria:

* Must have spoken to a healthcare provider about treatment for depression in the past 12 months
* Must have started or stopped medication for depression between January 2018 and their surveyed date.

Exclusion Criteria:

* None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample of adults in the United States who have made decision about treatment of depression in the past 12 months will be recruited from an online panel.
Sampling Method: Non-Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will create a complete, cleaned, de-identified copy of the final data set for each online field test.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will be available to outside investigators starting 6 months after publication.
Access Criteria: Information about the data sets will be on the Health Decision Sciences Center website and in publications of the data. Dr. Sepucha will share a de-identified data set with outside investigators at no cost, according to approved Massachusetts General Hospital (MGH)/Partners policies for data sharing. Investigators from other sites will be able to request the data and will be required to complete a data use agreement that ensures that all local Institutional Review Board (IRB) requirements are met before using the data, that they will not attempt to identify any data in the dataset, and that they will not share the data set with anyone outside their project team.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: April 2020 - May 2020 using a national, non-probability panel obtained from Marketing Systems Group (MSG). MSG recruited participants by sending out invitation emails to potential responders.
Pre-assignment Details: Eligible respondents were adults in the US who had talked with a healthcare provider about starting or stopping medication for depression in the past 12 months. The sample was selected to have approximately equal age distribution above and below 40 years old (e.g. 18-39 and 40-75). Respondents were re-contacted approximately one-week post survey for a re-test survey.
Period: Overall Study
Arm/Group | Original Shared Decision Making Process Scale | Revised Shared Decision Making Process Scale
Started | 230 | 264
Completed | 230 | 264
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Web-based non-probability panel of respondents aged 18-75 years old who had discussed with their healthcare provider about starting or stopping treatment for depression in the past year. Participants needed to have provided enough information to calculate the shared decision making process score (primary outcome of interest)
Groups:
- Total: Total of all reporting groups
Arm/Group | Original Shared Decision Making Process Scale | Revised Shared Decision Making Process Scale | Total
Number analyzed (Participants) | 230 | 264 | 494
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (14) | 44 (14) | 43 (14)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 158 | 197 | 355
  Male | 72 | 66 | 138
  Non-Binary | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 23 | 35
  Not Hispanic or Latino | 218 | 241 | 459
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 8 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 14 | 26
  White | 193 | 224 | 417
  More than one race | 5 | 8 | 13
  Unknown or Not Reported | 10 | 11 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 230 | 264 | 494

OUTCOME MEASURES:

1. Primary Outcome: Shared Decision Making Process Score
Description: The Shared Decision Making Process is a short patient-reported survey that measures the amount of shared decision making that occurs in an interaction. Scores for both versions of the scale range from 0-4 where higher values indicate a better shared decision making process occurred.
Time Frame: Baseline survey
Population: participants who answered the shared decision making process items and provided sufficient information to calculate a SDM Process score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Original Shared Decision Making Process Scale | Revised Shared Decision Making Process Scale
Number analyzed (Participants) | 230 | 264
score on a scale | 2.35 (1.11) | 2.51 (1.05)
Statistical Analysis 1: Comparison: Original Shared Decision Making Process Scale vs Revised Shared Decision Making Process Scale; SDM Process score distributions were compared to determine of the scores spanned the range of possible values, were normally distributed, had low rates of missing data, and whether there was indications of floor or ceiling effects. we conducted independent t-tests to determine if there were differences in SDM Process scores between the two versions; Test type: Other; p = 0.092, t-test, 2 sided; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.02 to 0.33]

2. Secondary Outcome: Decisional Conflict Tool (SURE)
Description: Measures decisional conflict, consists of 4 yes/no items. Scores range 0-4 where 0 indicates high decisional conflict, 4 indicates no decisional conflict, and scores less than or equal to 3 indicate decisional conflict. The measure is top-scored and we report the percentage of participants who scored a 4 ("no decisional conflict).
Time Frame: Baseline survey
Population: participants who completed all 4 items of the short decisional conflict scale. Only 485/494 participants provided enough information to calculate a SURE score.
Measure: Number; unit: percentage of patients
Arm/Group | Original Shared Decision Making Process Scale | Revised Shared Decision Making Process Scale
Number analyzed (Participants) | 227 | 258
percentage of patients | 63 | 72

3. Secondary Outcome: Decision Regret Scale
Description: 5-item decision regret scale ranges from 0-100 with higher scores indicating greater decisional regret.
Time Frame: Baseline survey
Population: Participants who answered all 5 decision regret questions. All 494 participants provided enough information to calculate decision regret score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Original Shared Decision Making Process Scale | Revised Shared Decision Making Process Scale
Number analyzed (Participants) | 230 | 264
score on a scale | 23 (18) | 21 (20)

4. Secondary Outcome: Single-Item Measure of Decision Regret
Description: Single item asking "If you knew then what you know now, do you think you would make the same decision about depression?" Responses are definitely yes, probably yes, probably no and definitely no.
Time Frame: Baseline survey
Population: participants who answered the single-item regret question.
Measure: Count of Participants; unit: Participants
Arm/Group | Original Shared Decision Making Process Scale | Revised Shared Decision Making Process Scale
Number analyzed (Participants) | 230 | 264
Participants
  Definitely yes | 119 | 134
  Probably yes | 95 | 102
  Probably no | 15 | 24
  Definitely no | 1 | 4

5. Secondary Outcome: Treatment Preference
Description: Single item asking "What did you want to do to manage your depression" with response options (1) Anti-depressant medicine alone, (2) Counseling or therapy alone, (3) Both medicine and counseling, and (4) Do something else.
Time Frame: Baseline survey
Population: participants who answered the treatment preference question. 493/494 provided information for this question
Measure: Count of Participants; unit: Participants
Arm/Group | Original Shared Decision Making Process Scale | Revised Shared Decision Making Process Scale
Number analyzed (Participants) | 230 | 263
Participants
  Anti-depressant medicine alone | 71 | 91
  Counseling or therapy alone | 28 | 28
  Both medicine and counseling | 125 | 138
  Do something else | 6 | 6

6. Secondary Outcome: Adapted Controlled Preference Scale
Description: Single item asking the participant who made the ultimate decision. The categorical response options are 1) the patient made the decision, 2)the provider made the decision, or 3) both patient and provider made the decision together.
Time Frame: Baseline survey
Population: participants who answered the controlled preference scale question.
Measure: Count of Participants; unit: Participants
Arm/Group | Original Shared Decision Making Process Scale | Revised Shared Decision Making Process Scale
Number analyzed (Participants) | 230 | 264
Participants
  Mainly my decision | 107 | 125
  Mainly the healthcare provider's decision | 32 | 27
  We made the decision together | 91 | 112

7. Secondary Outcome: Shared Decision Making Process Measure Retest
Description: The Shared Decision Making Process is a short patient-reported survey that measures the amount of shared decision making that occurs in an interaction. Scores range from 0-4 where higher values indicate a better shared decision making process occurred.
Time Frame: 1 week after baseline survey
Population: A subset of participants who completed the baseline survey (n=200) were re-contacted approximately 1 week post-survey for a retest. Participants who completed the retest survey and provided enough information to calculate the shared decision making process score were part of this analysis. 163/200 participants provided sufficient information to calculate a retest SDM Process score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Original Shared Decision Making Process Scale | Revised Shared Decision Making Process Scale
Number analyzed (Participants) | 79 | 84
score on a scale | 2.27 (1.05) | 2.58 (0.97)

8. Secondary Outcome: Depression Knowledge
Description: Multiple choice knowledge items for each topic will be combined to a total knowledge score (0-100) with higher scores indicating higher knowledge
Time Frame: Baseline survey
Population: participants who completed at least 60% of the knowledge questions for their respective cancer screening group. All 494 participants provided sufficient information to calculate a knowledge score.
Measure: Mean (Standard Deviation); unit: percentage of correct answers
Arm/Group | Original Shared Decision Making Process Scale | Revised Shared Decision Making Process Scale
Number analyzed (Participants) | 230 | 264
percentage of correct answers | 55.22 (22.96) | 55.98 (21.87)

9. Secondary Outcome: Adherence
Description: 3 item measure of adherence to medication for sample participants who indicate that they are taking medicine. A total score is calculated with scores ranging form 0-100; higher values indicated greater medication adherence.
Time Frame: Baseline survey
Population: participants who completed all 3 measures of adherence to calculate an adherence score. 373/494 provided sufficient information to calculate an adherence score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Original Shared Decision Making Process Scale | Revised Shared Decision Making Process Scale
Number analyzed (Participants) | 169 | 204
score on a scale | 83.6 (18.47) | 84.79 (18.25)

ADVERSE EVENTS:
Time Frame: Survey responses were assessed within 2 weeks of survey completion for evidence of adverse events.
Description: In addition to reviewing survey responses, participants were given the contact information for 3 members of the study team prior to the start of the survey should they experience a problem or need to report an adverse event.
Arm/Group | Original Shared Decision Making Process Scale | Revised Shared Decision Making Process Scale
All-Cause Mortality (participants affected / at risk) | 0/230 | 0/264
Serious Adverse Events (participants affected / at risk) | 0/230 | 0/264
Other Adverse Events (participants affected / at risk) | 0/230 | 0/264

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT04343534/Prot_SAP_000.pdf